CLINICAL TRIAL: NCT00641745
Title: Long-Term Safety, Tolerability, and Effectiveness of Lurasidone in Subjects With Schizophrenia or Schizoaffective Disorder: A Randomized, Active Comparator-Controlled Trial
Brief Title: Lurasidone HCl - A Long Term Safety Phase 3 Study of Patients With Clinically Stable Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1050237
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Results first posted 2011-10-06 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Lurasidone; Schizophrenia; Latuda
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Lurasidone Hydrochloride; Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Lurasidone
  Interventions: Drug: Lurasidone HCl
- 2 (Active Comparator): Risperidone
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Lurasidone HCl — 40 - 120mg per day
  Arms: 1
Drug: Risperidone — Risperidone
  Arms: 2

SUMMARY:
Lurasidone HCl is a compound being developed for the treatment of schizophrenia. This clinical study is designed to test the hypothesis that lurasidone is safe and tolerable long term among clinically stable patients. The study will also assess the long term effectiveness of lurasidone as compared to an active comparator.

ELIGIBILITY:
Main Inclusion Criteria:

To be eligible to enter the study, each patient must comply with the following inclusion criteria:

* Subject is 18 to 75 years on the day of signing the consent form (age parameters may be restricted further per local requirements without protocol amendment).
* Subject meets Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for a primary diagnosis of schizophrenia (including disorganized (295.10), paranoid (295.30), undifferentiated (295.90), catatonic (295.20), or residual (295.60) or schizoaffective disorder (295.70) subtypes.
* Subject is not pregnant or nursing, and is not planning pregnancy within the projected duration of the study.
* Subject will comply with the study procedures and outpatient visit requirements in the opinion of the investigator.
* Subject voluntarily agrees to participate in the study by giving written informed consent.

Main Exclusion Criteria:

To be excluded from entering this study if they fulfil any of the criteria below:

* Subject has a chronic organic disease of the central nervous system (other than schizophrenia).
* Subject has current clinically significant or history of, alcohol abuse/alcoholism or drug abuse/dependence within the last 6 months.
* In the opinion of the investigator, the subject has any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study.
* Subject has participated in a study with an investigational compound or device within 30 days of signing informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (73):
- United States (41):
  - K&S Professional Research Services LLC, Little Rock, Arkansas
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - South Coast Clinical Trials, Inc., Anaheim, California
  - Comprehensive NeuroScience, Inc. - Cerritos, Cerritos, California
  - Clinical Innovations Inc., Costa Mesa, California
  - Collaborative Neuroscience Network Inc, Garden Grove, California
  - University of Southern California, Los Angeles, California
  - Excell Research, Oceanside, California
  - University of California at Irvine Medical Center, Orange, California
  - Pasadena Research Institute, Pasadena, California
  - CNRI-Los Angeles, LLC, Pico Rivera, California
  - Clinical Innovations Inc., Riverside, California
  - CNRI-San Diego LLC, San Diego, California
  - UCSD, Outpatient Psychiatric Services, San Diego, California
  - Clinical Innovations Inc., Santa Ana, California
  - Collaborative Neuroscience Network Inc, Torrance, California
  - Comprehensive NeuroScience, Inc., Washington D.C., District of Columbia
  - Fidelity Clinical Research Inc., c/o Segal Institute for Clinical Research, North Miami, Florida
  - Fidelity Clinical Research Inc., North Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Northlake Medical Research Center, Tucker, Georgia
  - Alexian Brothers Medical Center, Hoffman Estates, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Precise Research Center, Flowood, Mississippi
  - St. Charles Psychiatric Associates - Midwest Research, Saint Charles, Missouri
  - St. Louis Clinical Trials, St Louis, Missouri
  - Creighton University, Omaha, Nebraska
  - CRI Worldwide, Willingboro, New Jersey
  - SUNY Downstate University, Brooklyn, New York
  - Neurobehavioral Research Inc., Cedarhurst, New York
  - Manhattan Psychiatric Center, New York, New York
  - Social Psychiatry Research Institute, New York, New York
  - University of North Carolina at Chapel Hill, Raleigh, North Carolina
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Research Strategies of Memphis LLC, Memphis, Tennessee
  - Community Clinical Research, Inc., Austin, Texas
  - Pillar Clinical Research LLC, Dallas, Texas
  - Claghorn-Lesem Research Clinic, Inc., Houston, Texas
  - Alliance Research Group, Richmond, Virginia
- Argentina (5):
  - Fundación para el Estudio y Tratamiento de las Enf. Mentales, Capital Federal, BUE
  - Clinica Privada Neuropsiquiatrica San Agustin, La Plata, BUE
  - Resolution Psychopharmacology Research Institute, Mendoza, MEN
  - CIAP, Rosario, SFE
  - Sanatorio 'Prof. Leon S. Morra' S.A., Córdoba
- Brazil (4):
  - Sanatorio Sao Paulo, Salvador, Estado de Bahia
  - Hospital Espirita de Psiquiatria Bom Retiro, Curitiba, Paraná
  - Hospital Mario Kroeff, Rio de Janeiro, Rio de Janeiro
  - PAX Clinica Psiquiatrica Ltda, Aparecida de Goiânia
- Chile (5):
  - Hospital Clincio Felix Bulnes, Quinta Normal, Santiago Metropolitan
  - Instituto Psiquiátrico Dr. José Horwitz Barak, Recoleta, Santiago Metropolitan
  - Hospital Barros Luco Trudeau, San Miguel, Santiago Metropolitan
  - CIPAM - Clínica Pedro Montt, Santiago, Santiago Metropolitan
  - Hospital Base Valdivia, Valdivia, Valdivia
- Croatia (3):
  - Psychiatric Hospital Vrapce, Zagreb, City of Zagreb
  - Croatian institute for brain research Neuron, Zagreb, City of Zagreb
  - Clinical Hospital Centre Rijeka, Rijeka, Rijeka
- Israel (5):
  - Beer Ya'acov Mental Health Center, Beer Yaakov, Beer Yaakov
  - Rambam Health Care Campus, Haifa, Haifa District
  - Shalvata Mental Health Center, Hod HaSharon, Hod Hasharon
  - Chaim Sheba Medical Center, Ramat Gan, Ramat Gan
  - Shalvata Mental Health Center, Ward B, Hod HaSharon
- South Africa (7):
  - Oranje Hospital, Bloemfontein, Free State
  - Rand Clinic, Johannesburg, Gauteng
  - Private Practice, Pretoria, Gauteng
  - Flexivest fourteen Research Centre, Cape Town, W Cape
  - Cape Trial Centre, Cape Town
  - Crompton Medical Centre East, Natal
  - Weskoppies Hospital, Pretoria West
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Chulalongkorn University, Bangkok
  - Somdet Chaopraya Institute of Psychiatry, Klongsan, Bangkok
  - Suan Prung Psychiatric Hospital, Muang, Chiang Mai

REFERENCES:
- [Background] Keefe RS, Fox KH, Harvey PD, Cucchiaro J, Siu C, Loebel A. Characteristics of the MATRICS Consensus Cognitive Battery in a 29-site antipsychotic schizophrenia clinical trial. Schizophr Res. 2011 Feb;125(2-3):161-8. doi: 10.1016/j.schres.2010.09.015. Epub 2010 Dec 31. PMID 21075600
- [Result] Citrome L, Cucchiaro J, Sarma K, Phillips D, Silva R, Tsuchiya S, Loebel A. Long-term safety and tolerability of lurasidone in schizophrenia: a 12-month, double-blind, active-controlled study. Int Clin Psychopharmacol. 2012 May;27(3):165-76. doi: 10.1097/YIC.0b013e32835281ef. PMID 22395527
- [Derived] Patel PJ, Weidenfeller C, Jones AP, Nilsson J, Hsu J. Long-Term Assessment of Lurasidone in Schizophrenia: Post Hoc Analysis of a 12-Month, Double Blind, Active-Controlled Trial and 6-Month Open-Label Extension Study. Neurol Ther. 2021 Jun;10(1):121-147. doi: 10.1007/s40120-020-00221-4. Epub 2020 Oct 24. PMID 33098548
- [Derived] Mattingly GW, Haddad PM, Tocco M, Xu J, Phillips D, Pikalov A, Loebel A. Switching to Lurasidone following 12 months of treatment with Risperidone: results of a 6-month, open-label study. BMC Psychiatry. 2020 May 5;20(1):199. doi: 10.1186/s12888-020-02523-1. PMID 32370778
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500

RESULTS

PARTICIPANT FLOW:
Groups:
- Lurasidone: Lurasidone 40 mg tablets (flexibly dosed): 40-120 mg/day
- Risperidone: Risperidone 2 mg tablets (2-6 mg/day) flexibly dosed
Period: Overall Study
Arm/Group | Lurasidone | Risperidone
Started | 427 | 202
Completed | 147 | 89
Not Completed | 280 | 113

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone | Risperidone | Total
Number analyzed (Participants) | 427 | 202 | 629
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (11.3) | 41.6 (11.3) | 41.7 (11.3)
Gender [Number; unit: participants] — There were 9 subjects randomized to lurasidone but did not take study drug and thus there is a discrepancy of 9 subjects in the lurasidone treatment group between the participant population and the overall number of baseline participants.
  participants
    Female | 117 | 76 | 193
    Male | 302 | 126 | 428
Region of Enrollment [Number; unit: participants] — There were 9 subjects randomized to lurasidone but did not take study drug and thus there is a discrepancy of 9 subjects in the lurasidone treatment group between the participant population and the overall number of baseline participants.
  participants
    United States | 279 | 133 | 412
    Argentina | 24 | 13 | 37
    Brazil | 15 | 9 | 24
    Thailand | 13 | 3 | 16
    Croatia | 7 | 5 | 12
    Israel | 3 | 0 | 3
    Chile | 19 | 7 | 26
    South Africa | 59 | 32 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Lurasidone | Risperidone
Number analyzed (Participants) | 427 | 202
participants | 395 | 189

ADVERSE EVENTS:
Time Frame: 14 days post-study therapy
Arm/Group | Lurasidone | Risperidone
Serious Adverse Events (participants affected / at risk) | 46/419 | 20/202
Other Adverse Events (participants affected / at risk) | 349/419 | 169/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=419) | Risperidone (N=202)
Hypertensive Heart Disease (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Oculogyric Crisis (Eye disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forearm Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Antepartum Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Conduct Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delusion of Reference (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 12 (12) | 8 (8)
Schizoaffective Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 8 (8) | 3 (3)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 2 (2)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Dsypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Physical Assault (Social circumstances) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=419) | Risperidone (N=202)
Constipation (Gastrointestinal disorders) | 8 (8) | 14 (14)
Nausea (Gastrointestinal disorders) | 70 (70) | 22 (22)
Vomiting (Gastrointestinal disorders) | 42 (42) | 7 (7)
Nasopharyngitis (Infections and infestations) | 22 (22) | 13 (13)
Weight Decreased (Investigations) | 31 (31) | 9 (9)
Weight Increased (Investigations) | 39 (39) | 40 (40)
Akathisia (Nervous system disorders) | 60 (60) | 16 (16)
Dizziness (Nervous system disorders) | 25 (25) | 8 (8)
Dystonia (Nervous system disorders) | 12 (12) | 11 (11)
Headache (Nervous system disorders) | 42 (42) | 30 (30)
Parkinsonism (Nervous system disorders) | 18 (18) | 11 (11)
Sedation (Nervous system disorders) | 61 (61) | 28 (28)
Somnolence (Nervous system disorders) | 57 (57) | 36 (36)
Anxiety (Psychiatric disorders) | 38 (38) | 17 (17)
Insomnia (Psychiatric disorders) | 66 (66) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No